CLINICAL TRIAL: NCT01741233
Title: The Genetics Behind Vitamin D Status (VitDgen)
Acronym: VitDgen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Lone Banke Rasmussen, M.Sc., Ph.D., Technical University of Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-4-2012-071
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2012-12

CONDITIONS: Vitamin D Deficiency
Keywords: SNPs; vitamin D; Vitamin D status; UVB irradiation; genetics
MeSH Terms: conditions — Vitamin D Deficiency

ARMS (1):
- UV-B irraditation (Experimental): VitDgen
  Interventions: Genetic: VitDgen

INTERVENTIONS:
Genetic: VitDgen

SUMMARY:
The overall purpose of the study is to investigate whether there is a relationship between 26 different single nucleotide polymorphisms (SNPs) in the vitamin D pathway, ultraviolet B (UV-B) irradiation of the skin and vitamin D status.

The hypothesis is that vitamin D status are influated by different genetic genotypes in the vitamin D pathway.

DETAILED DESCRIPTION:
In this study approximately 80 participants (over 18 years) are included. All the participants has previously participated in the VitmaD intervention study (NCT01184716) .

Participants will in total receive 4 times UV-B irradiation (3 SED) with two day apart each time, to stimulate vitamin D production in the skin. The participants skintype will be measured. The study starts in January 2013 and runs to the end of Marts 2013. During this winter period, it is in Denmark not possible to produce vitamin D in the skin through sunlight exposure.

ELIGIBILITY:
Inclusion Criteria:

* Health participants over 18 years, that previously participated in VitmaD intervention study

Exclusion Criteria:

* skindiseases
* intake of medicin that causes photosensitive skin
* pregnant or nursing
* sun vacation 3 month before the intervention
* intake of vitamin D supplement 3 month before the intervention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D | 10 days
  Measures the vitamin D status i serum at baseline and at the end of the project

SECONDARY OUTCOMES:
Skintest | 10 days
  Optimize scientific; measures pigmentation and redness of the skin. Are measured at baseline and at end of project

CONTACTS AND LOCATIONS:
Overall Officials: Lone Rasmussen, M.Sc., Ph.D., Principal Investigator — DTU, Denmark
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Bispebjerg, Copenhagen
  - DTU / National Food Institute, Mørkhøj, Søborg

REFERENCES:
- [Derived] Nissen J, Vogel U, Ravn-Haren G, Andersen EW, Madsen KH, Nexo BA, Andersen R, Mejborn H, Bjerrum PJ, Rasmussen LB, Wulf HC. Common variants in CYP2R1 and GC genes are both determinants of serum 25-hydroxyvitamin D concentrations after UVB irradiation and after consumption of vitamin D(3)-fortified bread and milk during winter in Denmark. Am J Clin Nutr. 2015 Jan;101(1):218-27. doi: 10.3945/ajcn.114.092148. Epub 2014 Nov 5. PMID 25527766